CLINICAL TRIAL: NCT03169140
Title: Effect of Biofreeze®, TheraBand® Kinesiology Tape, or the Combination of Products on Acute Low Back Pain, Disability, and Range of Motion
Brief Title: Effect of at Home Pain Management Products on Acute Low Back Pain, Disability, and Range of Motion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decided not to proceed
Sponsor: Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Low Back Home Care
Record Dates: First submitted 2017-05-16; First posted 2017-05-30 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Low Back Pain; Acute Pain
Keywords: pain management; topical analgesic; acute low back pain; kinesiology tape
MeSH Terms: conditions — Low Back Pain; Acute Pain; Agnosia | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Group 1 (Active Comparator): Receive a combination of products (TheraBand Kinesiology Tape and Biofreeze) to use for one week for at home pain management.
  Interventions: Device: TheraBand Kinesiology Tape; Device: Biofreeze
- Group 2 (Active Comparator): Receive TheraBand Kinesiology Tape product to use for one week for at home pain management.
  Interventions: Device: TheraBand Kinesiology Tape
- Group 3 (Active Comparator): Receive a topical product, Biofreeze, to use for one week for at home pain management
  Interventions: Device: Biofreeze
- Group 4 (Active Comparator): Receive advice sheet outlining at home pain management strategies to use for one week.
  Interventions: Behavioral: Advice

INTERVENTIONS:
Device: TheraBand Kinesiology Tape — A 20 cm strip of tape will be applied to each side of the low back directly over the erector spinae muscles at the site of pain. This tape will remain there, and be reapplied when necessary, for one week.
  Arms: Group 1; Group 2
Device: Biofreeze — The topical analgesic will be sprayed directly on top of the erector spinae and site of pain low back directly, from inferior to superior to inferior 4 times a day for one week.
  Arms: Group 1; Group 3
Behavioral: Advice — An at-home pain management care sheet, outlining standard care advice will be followed for at home pain management for one week.
  Arms: Group 4

SUMMARY:
The purpose of this study is to compare the effect of a combination of separate therapies of Biofreeze® and TheraBand Kinesiology Tape to advice on acute pain, disability and fear avoidance among low back patients over a 1-week period of time.

DETAILED DESCRIPTION:
A convenience sample of 120 acute low back pain patients will be recruited from Sport and Spine Rehab at their initial appointment. Exclusionary criteria will include pregnancy, cancer, or a corticosteroid injection within the past 2 weeks. Additionally, anyone who has a history of low back surgery will be excluded. Patients will be recruited following their initial examination if they meet the inclusion criteria of reporting low back pain for less than 2 weeks and be >18 years of age. Patients will complete the informed consent, demographics information questionnaire, Numeric Pain Rating Scale (NPRS), Roland-Morris Low Back Pain and Disability Questionnaire (RMDQ), Fear Avoidance Beliefs Questionnaire (FABQ). Following paper documents their lumbar range of motion and posture will be analyzed using the DorsaVi ViMove device [http://us.dorsavi.com/vimove/] (T1). After completing T1, patients will then be randomized into 1 of 4 at-home pain management groups (n=30 per group), to be followed for one week. Group 1 (Biofreeze® + Tape), Group 2 (Tape Only), Group 3 (Biofreeze Only), and Group 4 (Advice Alone). Treatment at the first office visit will be standardized to include manipulation only; no in-office therapy will be provided to either group at the first visit. Upon returning for their 2nd (T2), and 3rd (T3) office visits, all patients will rate their pain (NPRS). At one week (T4) patients will complete the paper and pencil instruments from the first visit, which assess the subjects' pain on the Numeric Pain Rating Scale (NPRS), low back disability on the Roland-Morris Low Back Pain and Disability Questionnaire (RMDQ), and fear on the Fear Avoidance Beliefs Questionnaire (FABQ). Lumbar range of motion and posture will also be reassessed. In addition,, at home pain management compliance and pain medication will be documented on a daily basis for the entire week.

ELIGIBILITY:
Inclusion Criteria:

* low back pain for less than 2 weeks and 18 years of age or older

Exclusion Criteria:

* pregnancy, cancer, or a corticosteroid injection within the past 2 weeks and a history of low back surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Numeric Pain Rating Scale (NPRS) over one week | Baseline (T1), Day 2 (T2), Day 4 (T3), 1 week (T4)
Change in Roland-Morris Low Back Pain and Disability Questionnaire (RMDQ) over one week | Baseline (T1), 1 week (T4)
Change in Fear Avoidance Beliefs Questionnaire (FABQ) over one week | Baseline (T1), 1 week (T4)
Change in lumbar range of motion over one week | Baseline (T1), 1 week (T4)
  Using the DorsaVi sensor technology lumbar flexion, extension, and side bending will be measures

CONTACTS AND LOCATIONS:
Locations (1):
- Sport and Spine Rehab, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No